CLINICAL TRIAL: NCT05097586
Title: Randomized Controlled Trial of At-home Transcranial Direct Current Stimulation (tDCS) for Depression in Pregnancy
Brief Title: RCT of At-Home tDCS for Depression in Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: Centre for Addiction and Mental Health (Other); Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Simone Vigod, Principal Investigator, Professor of Psychiatry, Senior Scientist, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTO Project ID: 3263
Record Dates: First submitted 2021-10-01; First posted 2021-10-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Major Depression; Pregnancy; Postpartum Depression
Keywords: Pregnancy; Depression; Transcranial direct current stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Depression, Postpartum; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active tDCS (Experimental): 2mA of direct current delivered to the dorsolateral prefrontal cortex for 30 minutes each, 5 times per week for 3 weeks, for a total of 15 sessions using the Soterix Medical tDCS mini-CT model 1601-LTE.
  Interventions: Device: active tDCS; Other: workbook
- control (Sham Comparator): Sham stimulation where the current is turned off after 30 seconds in a slow ramp down, delivered to the dorsolateral prefrontal cortex for 30 minutes each, 5 times per week for 3 weeks, for a total of 15 sessions using the Soterix Medical tDCS mini-CT model 1601-LTE.
  Interventions: Other: workbook; Device: sham tDCS

INTERVENTIONS:
Device: active tDCS — 2mA of direct current delivered in 15 sessions lasting 30 minutes each over 3 weeks
  Arms: active tDCS
Other: workbook — Self-directed depression in pregnancy workbook completed during each session to control the in-session brain state
Device: sham tDCS — Sham stimulation in which the current turns off after 30 seconds in a slow ramp down that mirrors sensory adaptation in ongoing stimulation, delivered in 15 sessions lasting 30 minutes each over 3 weeks
  Arms: control

SUMMARY:
This is a randomized, sham-controlled trial to determine whether treatment with transcranial direct current stimulation (tDCS) is superior to a sham condition at reducing the symptoms of depression in pregnant people with moderate to severe depression. The study aims to enrol 156 participants across all sites. Data collection occurs at baseline, immediately after treatment, every 4 weeks during pregnancy and 4-, 12-, 26- and 52-weeks postpartum

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) is a brain stimulation technique for the treatment of depression that has great potential for filling the gap in treatment options for moderate and severe depression in pregnancy. Participants are randomized 1:1 to active tDCS treatment or sham control. After at least one in-person training session with the research team, participants take the tDCS device home and self-administer 30-minute treatments 5 times per week, for 3 weeks, for a total of 15 sessions. Rater-administered and self-report outcomes are collected weekly during the 3-week active treatment phase, every 4 weeks during pregnancy, and at 4-, 12-, 26- and 52-weeks postpartum. A mixed methods process evaluation is embedded into the trial.

ELIGIBILITY:
Inclusion criteria:

1. Adult, ≥18 years of age
2. Singleton pregnancy, 12 to end of 32 weeks single gestation at randomization
3. In a major depressive episode (MDE) with at least moderate symptom severity (PHQ-9 ≥10 and confirmed using MINI International Neuropsychiatric Interview as MDE without psychotic features)
4. Assessed by a psychiatrist at one of the study recruitment sites during pregnancy, and offered the option of antidepressant medication for treatment but declined to use
5. No new treatments for depression (i.e. psychological or somatic) and no pharmacological treatment for depression in the 4 weeks prior to starting treatment

Exclusion criteria:

1. Active alcohol or substance use disorder in previous 12 months as assessed by GAIN-SS
2. Active suicidality as assessed by the Columbia Suicide Severity Rating Scale (C-SSRS)
3. Bipolar disorder as assessed by MINI International Neuropsychiatric Interview
4. Schizophrenia or other psychotic disorder as assessed by MINI International Neuropsychiatric Interview
5. Major unstable or life-threatening medical illness (e.g. such as advanced cancer), pre-eclampsia/eclampsia in current pregnancy or neurologic illness or seizure history
6. Major congenital anomalies or major obstetrical complications in current pregnancy (determined by clinical PI/Co-I assessment)
7. Metal implants in cranium or any electrical implants
8. Benzodiazepine (except intermittent low-dose lorazepam no more than 2mg equivalent per day) or anticonvulsant use as these interfere with anodal tDCS
9. Visibly non-intact skin/rash on scalp areas at stimulation electrode sites
10. Unable to consent or complete study measures in English, or unable to complete depression in pregnancy workbook (the attention-control) in French or English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms post treatment | End of Week 3 of treatment
  Depressive symptoms are measured with the 10-item rater-administered Montgomery Asberg Depression Rating Scale (MADRS).The MADRS is a standard rater-administered measure with good reliability and validity in clinical populations; interviewers can achieve and maintain high levels of inter-rater reliability. Nine items are based upon patient report and one on rater observation. Items are rated on a 0-6 continuum (0=no abnormality, 6=severe; score range 0-60). A MADRS score of <11 indicates remission

SECONDARY OUTCOMES:
Remission of depression | 4 weeks postpartum
  Measured with the 10-item rater-administered Montgomery Asberg Depression Rating Scale (MADRS).The MADRS is a standard rater-administered measure with good reliability and validity in clinical populations; interviewers can achieve and maintain high levels of inter-rater reliability. Nine items are based upon patient report and one on rater observation. Items are rated on a 0-6 continuum (0=no abnormality, 6=severe; score range 0-60). A MADRS score of <11 indicates remission
Depressive symptoms | End of Week 1, and Week 2 of treatment, q4 weeks during pregnancy, and 4-, 12-, 26- and 52-weeks postpartum
  measured with the 10-item rater-administered Montgomery Asberg Depression Rating Scale (MADRS).The MADRS is a standard rater-administered measure with good reliability and validity in clinical populations; interviewers can achieve and maintain high levels of inter-rater reliability. Nine items are based upon patient report and one on rater observation. Items are rated on a 0-6 continuum (0=no abnormality, 6=severe; score range 0-60). A lower score indicates less severe symptoms.
Self-reported depressive symptoms | End of Week 1, Week 2 and Week 3 of treatment, q4 weeks during pregnancy (up to 28 weeks), and 4-, 12-, 26- and 52-weeks postpartum (up to 80 weeks)
  Depressive symptoms will be measured using the Edinburgh Postnatal Depressive Scale (EPDS), a self-report scale that has been validated for use in pregnancy and postpartum. EPDS scores range from 0 to 30. EPDS scores >12 are predictive of a diagnosis of depression, with higher scores indicating more severe symptoms
Self-reported anxiety symptoms | End of Week 1, Week 2 and Week 3 of treatment, q4 weeks during pregnancy (up to 28 weeks), and 4-, 12-, 26- and 52-weeks postpartum (up to 80 weeks)
  Measured using the Generalized Anxiety Disorder-7 (GAD-7) scale which is a self-report scale with good discriminate validity in perinatal populations. GAD-7 scores range from 0 to 21, with higher scores indicating more severe symptoms
Maternal Quality of Life (QoL) | End of Week 1, Week 2 and Week 3 of treatment, q4 weeks during pregnancy (up to 28 weeks), and 4-, 12-, 26- and 52-weeks postpartum (up to 80 weeks)
  Measured using 12-Item Short Form Survey (SF-12), a 12-item measure often used to estimate quality-adjusted life year (QALY), a preference-based utility measure of health-related QoL as perceived by the patient and the gold standard measure of effectiveness recommended for economic evaluation. SF12 scores consist of Physical and Mental Component Summaries. Scores range from 0-100 with higher scores indicating better functioning
Health Service Use: Health System Costs | End of Week 3 of treatment, q4 weeks during pregnancy (up to 28 weeks), and 4-, 12-, 26- and 52-weeks postpartum (up to 80 weeks)
  Calculated from participant self-report of medical costs such as hospitalization, visits with health professionals and medications
Health Service Use: Productivity Loss | End of Week 3 of treatment, q4 weeks during pregnancy (up to 28 weeks), and 4-, 12-, 26- and 52-weeks postpartum (up to 80 weeks)
  Calculated from participant self-report of activities and time commitment related to attending appointments and obtaining services, work absences of the patient and family members
Health Service Use: Participant Cost | End of Week 3 of treatment, q4 weeks during pregnancy (up to 28 weeks), and 4-, 12-, 26- and 52-weeks postpartum (up to 80 weeks)
  Calculated from participant self-report of costs related to attending appointments and obtaining services
Dyadic Relationship | End of Week 3 of treatment, q4 weeks during pregnancy (up to 28 weeks), and 4-, 12-, 26- and 52-weeks postpartum (up to 80 weeks)
  Relationship satisfaction measured using the Dyadic Consensus Subscale, a 13-item subscale of the 32-item Dyadic Adjustment Scale (DAS). This self-report measure of the extent of agreement between partners is valid for measuring overall dyadic adjustment. Higher scores indicate a higher degree of dyadic consensus
Maternal Birth Outcomes | End of Week 1, Week 2 and Week 3 of treatment, q4 weeks during pregnancy (up to 28 weeks), and 4 weeks postpartum (up to 32 weeks)
  Self-reported pregnancy and birth complications querying indicators recommended by the Canadian Perinatal Surveillance System (CPSS)
Neonatal Birth Outcomes | 4 weeks postpartum (up to 32 weeks)
  Self-reported neonatal birth outcomes including medical conditions and complications querying indicators recommended by the Canadian Perinatal Surveillance System (CPSS)
Maternal Child Relationship | 4-, 12-, 26- and 52-weeks postpartum (up to 80 weeks)
  Parenting stress is measured by the Parenting Stress Index Short Form (PSI-SF) which is a 36-item measure consisting of 6 sub-scales: parental distress, dysfunction in the parent-child relations and difficult child. Scores range from 36 to 180. Higher scores indicate higher levels of parenting stress
Infant Temperament | 12 and 52 weeks postpartum (up to 80 weeks)
  Measured using the Infant Characteristics Questionnaire (ICQ). The ICQ is a 27-item questionnaire with each item coded 1-7. Higher scores indicate higher parental perceptions of difficult infant temperament
Child Development | 12 and 52 weeks postpartum (up to 80 weeks)
  Assessed using the Ages and Stages Questionnaire (ASQ-3), a 30-item instrument that screens for child development from 1 to 60 months

OTHER OUTCOMES:
Concurrent Health Service Use | End of Week 1, Week 2 and Week 3 of treatment, q4 weeks during pregnancy (up to 28 weeks), and 4-, 12-, 26- and 52-weeks postpartum (up to 80 weeks)
  Self-reported concurrent mental health service use such as psychotherapy or antidepressant use that could confound treatment
Tolerability of Intervention | End of Week 1, Week 2 and Week 3 of treatment
  Assessed using the rater-administered Toronto Side Effects Scale which is an anti-depressant side effects scale
Stanford Expectancy Scale | Baseline
  Assesses participant expectations of treatment effectiveness
Integrity of Treatment Blindness Questionnaire | End of session 1, End of Week 3 of treatment
  Participants report whether they believe they have received the treatment or the sham control.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Grigoriadis, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Centre; Daniel Blumberger, MD, MSc, Principal Investigator — Centre for Addiction and Mental Health; Simone Vigod, MD, MSc, Principal Investigator — Women's College Hospital
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario